CLINICAL TRIAL: NCT06533332
Title: A First-in-Human, Phase 1 Safety, Tolerability, Pharmacokinetic, and Preliminary Efficacy Study of Escalating Doses of ERX-315 in Participants With Advanced Solid Tumors
Brief Title: A Phase 1 Trial of ERX-315 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EtiraRx Australia Pty Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERX-315-101
Record Dates: First submitted 2024-07-22; First posted 2024-08-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor; Metastatic Breast Cancer; Metastatic Ovarian Cancer; Metastatic Endometrial Cancer; Metastatic Liver Cancer; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Liver Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ERX-315 (Experimental): Active investigational therapy
  Interventions: Drug: ERX-315

INTERVENTIONS:
Drug: ERX-315 — Drug administered intravenously twice a week at increasing dose levels, with starting dose of 0.4mg/kg.

SUMMARY:
This is a Phase 1 study to assess the safety of ERX-315 in patients with advanced solid tumors that have failed approved systemic therapies.

DETAILED DESCRIPTION:
The goal of this open-label, dose escalation and cohort expansion Phase 1 clinical trial is to determine the safety, tolerability and pharmacokinetics of ERX-315 in patients with advanced solid tumors, who have progressed on prior approved systemic therapies. Participants will receive ERX-315 as an intravenous (IV) injection twice a week, over 21-day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age at the time of signing the informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patients must have histologically or cytologically confirmed solid tumor, primarily including but not limited to breast, ovarian, pancreatic, endometrial and hepatocellular carcinoma, that is advanced unresectable and/or metastatic disease for whom standard therapies do not exist or are no longer effective
* Patients must have measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Adequate baseline organ function and hematologic function
* Life expectancy >3 months

Exclusion Criteria:

* Systemic anti cancer therapy within 4 weeks of first dose of study drug
* Major surgery (as defined by the Investigator) within 4 weeks of first dose of study drug.
* Uncontrolled intercurrent illnesses
* Known history of LIPA deficiency, such as Wolman disease or Cholesterol ester storage disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities of ERX-315 | 21 days
  First cycle dose limiting toxicities characterized by type, frequency, severity, timing, seriousness, and relationship to study drug
Incidence of Adverse Events as a measure of safety and tolerability of ERX-315 | 84 days
  Adverse events as characterized by type, frequency, severity (grade), timing, seriousness, and relationship to study drug.
Incidence of laboratory abnormalities as a measure of safety and tolerability of ERX-315 | 84 days
  Laboratory abnormalities as characterized by type, frequency, severity, and timing.
Determination of the recommended phase 2 dose | 84 days
  To determine the recommended phase 2 dose(s) for additional evaluation of ERX-315 in clinical trials for participants with advanced solid tumors

SECONDARY OUTCOMES:
Assessment of pharmacokinetic outcome measure of Area under the plasma concentration versus time curve (AUC). | 21 days
  AUC will be determined by non-compartmental analysis and assessed after single and multiple doses of drug
Assessment of pharmacokinetic outcome measure of Peak Plasma concentration (Cmax) | 21 days
  Cmax will be determined by non-compartmental analysis and assessed after single and multiple doses of drug
Assessment of pharmacokinetic outcome measure of drug half-life (t1/2) | 21 days
  t1/2 will be assessed after single and multiple doses of drug
Antitumor activity of ERX-315 based on Objective response rate (ORR) | 84 days
  ORR will be assessed by RECIST v1.1
Antitumor activity of ERX-315 based on Best Overall Clinical Response (BOCR) | 84 days
  BOCR will be assessed by RECIST v1.1
Antitumor activity of ERX-315 based on Duration of response (DOR) | 84 days
  DOR will be assessed by RECIST v1.1 and time frame of response
Antitumor activity of ERX-315 based on Progression-free survival (PFS) | 84 days
  PFS will be assessed by RECIST v1.1 and time frame of response

OTHER OUTCOMES:
Impact on patient reported symptoms using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) Questionnaire | 84 days
  Effect of ERX-315 on the changes from baseline in patient reported symptoms using the PRO-CTCAE Questionnaire
Serum LIPA lipase activity as pharmacodynamic markers of ERX-315 activity | 84 days
  The effect of ERX-315 on serum LIPA lipase activity may be evaluated
Circulating tumor DNA levels as pharmacodynamic markers of ERX-315 activity | 84 days
  The effect of ERX-315 on circulating tumor DNA levels may be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Cosman, MBBS, Principal Investigator — The Kinghorn Cancer Centre
Locations (4):
- Australia (4):
  - Macquarie University Health, Ryde, New South Wales
  - The Kinghorn Cancer Center, Sydney, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - Icon Cancer Centre Adelaide, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No